CLINICAL TRIAL: NCT03006991
Title: Individual Study of Methotrexate Based on Pharmacogenomics and Pharmacometrics
Brief Title: Study of Methotrexate Given to Juvenile Idiopathic Arthritis Patients Based on Pharmacogenomics and Pharmacometrics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Mo Xiaolan, Mo Xiaolan, Guangzhou Women and Children's Medical Center
Other Study IDs: 81603203
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: methotrexate, Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA is extracted and stored in freezer with -80°C.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- good efficacy: using therapeutic drug monitoring to adjust the dose of methotrexate. patients can reach effective outcome.
  Interventions: Other: therapeutic drug monitoring
- poor efficacy: patients can not reach effective outcome.

INTERVENTIONS:
Other: therapeutic drug monitoring — dose of methotrexate can be adjusted by therapeutic drug monitoring.
  Groups: good efficacy

SUMMARY:
This study will integrate Pharmacogenomics and Pharmacometrics, to explore an effective concentration of MTXPGn for JIA pediatric patients, and set up a Population Pharmacokinetics model to provide reference for individual administration on JIA pediatric patients.

DETAILED DESCRIPTION:
In order to find out "The critical reasons for individual variances in MTX of JIA pediatric patients and quantize the influence of these factors", based on early research, this study will integrate Pharmacogenomics and Pharmacometrics, to explore an effective concentration of MTXPGn for JIA pediatric patients, and set up a Population Pharmacokinetics model to provide reference for individual administration on JIA pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with Juvenile Idiopathic Arthritis
* 7.5-10mg/m2 per week per dose of methotrexate
* all patients have been treated with methotrexate at least for 3 months

Exclusion Criteria:

* co-treated other drugs which can interact with methotrexate

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with Juvenile Idiopathic Arthritis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Genotypes as measured by polymerase chain reaction-restriction fragment length polymorphism | 3 months
  genotype are collected from hospital system.

SECONDARY OUTCOMES:
Concentration as measured by liquid chromatography mass spectrometry | 3 months
  concentration of methotrexate are collected from hospital system

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Mo, master, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guandong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yanagimachi M, Naruto T, Hara T, Kikuchi M, Hara R, Miyamae T, Imagawa T, Mori M, Kaneko T, Morita S, Goto H, Yokota S. Influence of polymorphisms within the methotrexate pathway genes on the toxicity and efficacy of methotrexate in patients with juvenile idiopathic arthritis. Br J Clin Pharmacol. 2011 Feb;71(2):237-43. doi: 10.1111/j.1365-2125.2010.03814.x. PMID 21219404
- See also: Influence of polymorphisms within the methotrexate pathway genes on the toxicity and efficacy of methotrexate in patients with juvenile idiopathic arthritis — http://www.ncbi.nlm.nih.gov/pubmed/?term=Influence+of+polymorphisms+within+the+methotrexate+pathway+genes+on+the+toxicity+and+efficacy+of+methotrexate+in+patients+with+juvenile+idiopathic+arthritis